CLINICAL TRIAL: NCT01849107
Title: Plasma Citrulline: A Marker for Monitoring & Quantifying Radiation-Induced Small Bowel Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young Seok Kim, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTR_SB_2013
Record Dates: First submitted 2013-04-28; First posted 2013-05-08 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Diarrhea; Anorexia; Dyspepsia
Keywords: Radiation-induced small bowel toxicity; Plasma citrulline
MeSH Terms: conditions — Diarrhea; Anorexia; Dyspepsia

ARMS (1):
- Plasma citrulline (Experimental)
  Interventions: Biological: Plasma citrulline

INTERVENTIONS:
Biological: Plasma citrulline

SUMMARY:
Small bowel irradiation results in epithelial cell loss and consequently impairs function and metabolism. A metabolic end product of small bowel enterocytes is plasma citrulline. The investigators evaluate the correlation between plasma citrulline level, dose-volume histogram of small bowel, and small bowel toxicity grade by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE ver.4.0) to investigate whether citrulline can be used as a biomarker for quantifying radiation-induced epithelial cell loss.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer patients
* Appropriate liver, renal, and bone marrow function for radiotherapy
* Willing to provide informed written consent
* At least 20 years old

Exclusion Criteria:

* prior abdominopelvic radiation therapy or chemotherapy or abdominal surgery
* Any contraindication to radiotherapy (i.e. Severe connective tissue disorder, etc.)
* Prior or simultaneous history of other malignancy
* On medication for small bowel disease or CTCAE 4.0 Grade 1 or higher toxicity before radiation
* Any treatment delay more than 1 week during radiotherapy
* No radiotherapy due to any other reason except small bowel toxicity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Serial changes in plasma citrulline level baseline, on 3rd week during, on the day of completion of radiotherapy, and 3 months post-radiotherapy. | 1 year

SECONDARY OUTCOMES:
Correlation coefficient between plasma citrulline and dose-volume histogram of small bowel. | 1 year

OTHER OUTCOMES:
Correlation coefficient between plasma citrulline and toxicity grade by CTCAE 4.0 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Atahan IL, Onal C, Ozyar E, Yiliz F, Selek U, Kose F. Long-term outcome and prognostic factors in patients with cervical carcinoma: a retrospective study. Int J Gynecol Cancer. 2007 Jul-Aug;17(4):833-42. doi: 10.1111/j.1525-1438.2007.00895.x. Epub 2007 Mar 15. PMID 17367320
- [Background] Letschert JG, Lebesque JV, Aleman BM, Bosset JF, Horiot JC, Bartelink H, Cionini L, Hamers JP, Leer JW, van Glabbeke M. The volume effect in radiation-related late small bowel complications: results of a clinical study of the EORTC Radiotherapy Cooperative Group in patients treated for rectal carcinoma. Radiother Oncol. 1994 Aug;32(2):116-23. doi: 10.1016/0167-8140(94)90097-3. PMID 7972904
- [Background] Crenn P, Vahedi K, Lavergne-Slove A, Cynober L, Matuchansky C, Messing B. Plasma citrulline: A marker of enterocyte mass in villous atrophy-associated small bowel disease. Gastroenterology. 2003 May;124(5):1210-9. doi: 10.1016/s0016-5085(03)00170-7. PMID 12730862
- [Background] Lutgens LC, Deutz NE, Gueulette J, Cleutjens JP, Berger MP, Wouters BG, von Meyenfeldt MF, Lambin P. Citrulline: a physiologic marker enabling quantitation and monitoring of epithelial radiation-induced small bowel damage. Int J Radiat Oncol Biol Phys. 2003 Nov 15;57(4):1067-74. doi: 10.1016/s0360-3016(03)00781-8. PMID 14575838
- [Background] Crenn P, Messing B, Cynober L. Citrulline as a biomarker of intestinal failure due to enterocyte mass reduction. Clin Nutr. 2008 Jun;27(3):328-39. doi: 10.1016/j.clnu.2008.02.005. Epub 2008 Apr 28. PMID 18440672
- [Background] Herbers AH, Feuth T, Donnelly JP, Blijlevens NM. Citrulline-based assessment score: first choice for measuring and monitoring intestinal failure after high-dose chemotherapy. Ann Oncol. 2010 Aug;21(8):1706-1711. doi: 10.1093/annonc/mdp596. Epub 2010 Jan 20. PMID 20089560
- [Background] Lutgens LC, Blijlevens NM, Deutz NE, Donnelly JP, Lambin P, de Pauw BE. Monitoring myeloablative therapy-induced small bowel toxicity by serum citrulline concentration: a comparison with sugar permeability tests. Cancer. 2005 Jan 1;103(1):191-9. doi: 10.1002/cncr.20733. PMID 15573372
- [Background] Packey CD, Ciorba MA. Microbial influences on the small intestinal response to radiation injury. Curr Opin Gastroenterol. 2010 Mar;26(2):88-94. doi: 10.1097/MOG.0b013e3283361927. PMID 20040865
- [Background] Lutgens LC, Deutz N, Granzier-Peeters M, Beets-Tan R, De Ruysscher D, Gueulette J, Cleutjens J, Berger M, Wouters B, von Meyenfeldt M, Lambin P. Plasma citrulline concentration: a surrogate end point for radiation-induced mucosal atrophy of the small bowel. A feasibility study in 23 patients. Int J Radiat Oncol Biol Phys. 2004 Sep 1;60(1):275-85. doi: 10.1016/j.ijrobp.2004.02.052. PMID 15337566
- [Background] Kim YS, Shin SS, Nam JH, Kim YT, Kim YM, Kim JH, Choi EK. Prospective randomized comparison of monthly fluorouracil and cisplatin versus weekly cisplatin concurrent with pelvic radiotherapy and high-dose rate brachytherapy for locally advanced cervical cancer. Gynecol Oncol. 2008 Jan;108(1):195-200. doi: 10.1016/j.ygyno.2007.09.022. Epub 2007 Oct 25. PMID 17963825
- [Background] Onal C, Kotek A, Unal B, Arslan G, Yavuz A, Topkan E, Yavuz M. Plasma citrulline levels predict intestinal toxicity in patients treated with pelvic radiotherapy. Acta Oncol. 2011 Nov;50(8):1167-74. doi: 10.3109/0284186X.2011.584557. Epub 2011 Aug 24. PMID 21864050
- [Background] Kim YS, Kim JH, Ahn SD, Lee SW, Shin SS, Nam JH, Kim YT, Kim YM, Kim JH, Choi EK. High-dose extended-field irradiation and high-dose-rate brachytherapy with concurrent chemotherapy for cervical cancer with positive para-aortic lymph nodes. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1522-8. doi: 10.1016/j.ijrobp.2008.10.024. Epub 2009 Feb 21. PMID 19231106
- [Background] Kim YS, Kim JH, Yoon SM, Choi EK, Ahn SD, Lee SW, Kim JC, Yu CS, Kim HC, Kim TW, Chang HM. lymph node ratio as a prognostic factor in patients with stage III rectal cancer treated with total mesorectal excision followed by chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):796-802. doi: 10.1016/j.ijrobp.2008.08.065. Epub 2009 Mar 14. PMID 19289261
- [Background] Lee YS, Kim YS, Kim JH, Ahn SD, Lee SW, Shin SS, Nam JH, Kim YT, Kim YM, Kim JH, Choi EK. Feasibility and outcome of concurrent chemoradiotherapy for recurrent cervical carcinoma after initial surgery. Tumori. 2010 Jul-Aug;96(4):553-9. doi: 10.1177/030089161009600407. PMID 20968134
- [Background] Park JH, Kim YS, Ahn SD, Choi EK, Shin SS, Kim YT, Kim YM, Kim JH, Yi SY, Nam JH. Concurrent chemoradiotherapy or radiotherapy alone for locally advanced cervical cancer in elderly women. Tumori. 2010 Nov-Dec;96(6):959-65. PMID 21388059
- [Background] Kim JY, Kim JY, Kim JH, Yoon MS, Kim J, Kim YS. Curative chemoradiotherapy in patients with stage IVB cervical cancer presenting with paraortic and left supraclavicular lymph node metastases. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):741-7. doi: 10.1016/j.ijrobp.2012.01.070. Epub 2012 Aug 14. PMID 22898382
- [Background] Kim YS, Park SH, Ahn SD, Lee JE, Choi EK, Lee SW, Shin SS, Yoon SM, Kim JH. Differences in abdominal organ movement between supine and prone positions measured using four-dimensional computed tomography. Radiother Oncol. 2007 Dec;85(3):424-8. doi: 10.1016/j.radonc.2007.10.031. Epub 2007 Nov 26. PMID 18036688
- [Background] Choi HJ, Kim YS, Lee SH, Lee YS, Park G, Jung JH, Cho BC, Park SH, Ahn H, Kim CS, Yi SY, Ahn SD. Inter- and intra-observer variability in contouring of the prostate gland on planning computed tomography and cone beam computed tomography. Acta Oncol. 2011 May;50(4):539-46. doi: 10.3109/0284186X.2011.562916. Epub 2011 Mar 10. PMID 21391773